CLINICAL TRIAL: NCT01160146
Title: Geisinger Education Intervention Study in Obesity Protocol
Acronym: GEISO
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009-0296
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Obesity
Keywords: Obestiy; Over weight; referral patterns; Continuing Medical Education
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle counseling: Clinicians provide lifestyle management counseling regarding healthful lifestyle behaviors and daily physical activity.
  1. Logging foods for accountability and counting calories
  2. Close attention to portion control and appropriate serving sizes of foods consumed
  3. Consumption of appropriate calorie and sugar free beverages
  4. Good meal distribution and avoidance of meal skipping
  5. Balance of food groups using the MyPlate concept (USDA Choose My Plate)-inclusion of all food groups with emphasis on fruits, vegetables, whole grains, low-fat dairy products and lean meat/fish/poultry
  6. Increasing physical activity with reasonable, sustainable exercise or activity. Working toward a goal of at least 30 minutes, 5 days per week

SUMMARY:
Overweight and obesity has become an epidemic which warrants more aggressive treatment. However, few primary care physicians (PCPs) address this issue or do not possess adequate education regarding treatment modalities such as nutrition counseling or bariatric surgery. The primary goal of this study will be to determine whether the referrals for weight management can be influenced through obesity education.

DETAILED DESCRIPTION:
Evaluation of educational interventions focusing on the treatment of obesity will include in person CME sessions, interactive game/virtual patient computer software and two 30 minute DVD/Web-based CME opportunities that the physicians can review at their leisure. These educational interventions were not completed as part of this research.

A control group will be comprised of those healthcare professionals who did not complete the CME survey.

Completion of the post education survey would be completed even if there was no study. The reward given to PCP's (free enrollment in CME session and either lab coat or $40 CME credit) was given for clinical purposes only and not for research. The study consists of the collection of PCP referral rates prior to the educational opportunity and then after the CME looking for a change to referral rates.

In June of 2009, an Obesity Educational Intervention Summit was attended by PCPs. This research seeks approval to perform data pulls consisting of referrals from their practice to the GI/Nutrition Clinic for potential bariatric surgery evaluation.

The information to be collected regarding the primary care providers' referral rates will be collected by a CDIS data pull by a data broker. The biostatistician will link survey responses to referral patterns and education type and will be true, only individual to have access to direct identifiers and in turn will provide PI and study team with de-identified summary data.

ELIGIBILITY:
Inclusion Criteria:

Geisinger General Internal and Family Medicine PCPs (include physician, physical assistants and CRNP):

* PCP must be active between May 2008 - May 2009
* Average patient age between 30-60 (no individual patients will be identified using personal identification)
* Minimum of 100 patients assigned to PC

Exclusion Criteria:

* PCPs from clinics/departments other than General Internal Medicine or Family Medicine will be excluded from the analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Geisinger's General Internal Medicine Primary Care Clinic Geisinger's Family Medicine Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Correlation of weight management referral rates and attitudes/barriers towards obesity | Referral rates are calculated over the course of one year
  Referral rates to a weight management clinic will be evaluated and correlated with clinicians attitudes towards treatment of obesity (as assessed by questionnaire).

SECONDARY OUTCOMES:
Change in referral rate by Continuing Medical Education and change in referral rate by clinician characteristic | Compare rates of referral in year prior to Continuing Medical Education versus one year after Continuing Medical Education and compare rates of referral in consecutive years
  Compare change in Weight Management clinic referral rates between clinicians that attend in-person Continuing Medical Education versus those that complete an innovative gaming system Continuing Medical Education versus those that complete a web-based Continuing Medical Education and evaluate the correlation between changing Weight Management clinic referral rates and clinician characteristics such as attitudes towards obesity, clinician age/gender, number of patients, age/gender of patients, and percent of patients that are obese.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Still, DO, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

REFERENCES:
- See also: Geisinger Health System — http://geisinger.org